CLINICAL TRIAL: NCT02195635
Title: A Phase 1, Open-label, Single-center, 2-period, Single Sequence Drug-drug Interaction Study to Evaluate the Effects of Octreotide Acetate Injection (Sandostatin®) on the Pharmacokinetics of Single-dose Telotristat Etiprate in Healthy Male and Female Subjects
Brief Title: Phase 1, Open-label, Drug-drug Interaction Study With Octreotide Acetate Injection and Telotristat Etiprate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-109-NRM; LX1606.109 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Drug Interactions
MeSH Terms: interventions — telotristat; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Experimental): Single oral dose of 500 mg telotristat etiprate on Day 1
  Interventions: Drug: Telotristat etiprate
- Period 2 (Other): Subcutaneous injections of 200 µg octreotide acetate three times daily with a single oral dose of 500 mg telotristat etiprate on Day 6
  Interventions: Drug: Telotristat etiprate; Drug: Octreotide acetate

INTERVENTIONS:
Drug: Telotristat etiprate — 500 mg telotristat etiprate
Drug: Octreotide acetate — 200 µg octreotide acetate three times daily
  Arms: Period 2

SUMMARY:
To evaluate the effect of octreotide acetate injections (200 µg 3 times daily [tid]) on the pharmacokinetics (PK) of telotristat ethyl and its metabolite LP-778902 relative to administration of single-dose telotristat etiprate in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females ≥18 to ≤55 years of age
* Body mass index 18.0 to 32.0 kg/m2, inclusive, at Screening
* Vital signs (after at least 5 minutes resting in a supine position) at Screening that are within the following ranges: Systolic blood pressure, 90 to 140 mm Hg; Diastolic blood pressure, 50 to 90 mm Hg; Heart rate 40 to 100 beats per minute (bpm)
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Able to comprehend and willing to sign an Informed Consent Form

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or electrocardiogram (ECG) findings at Screening or Check-in (Day 1) that, in the opinion of the Investigator and/or the Sponsor or Sponsor's representative, may interfere with any aspect of study conduct or interpretation of results
* Use of any medications (prescription or over-the-counter), herbal tea, energy drinks, herbal products (eg, St. John's Wort, garlic, milk thistle, etc.), or supplements/supratherapeutic doses of vitamins within 14 days prior to the first dose administration and throughout the duration of the study, with the exception of those approved by the Investigator and/or the Sponsor or Sponsor's representative
* Prior exposure to telotristat etiprate
* Use of tobacco, smoking cessation products, or products containing nicotine within 3 months prior to Screening and for the duration of the study
* History of any major surgery within 6 months prior to Screening
* History of renal disease
* History of hepatic disease, or significantly abnormal liver function tests (>1.5 x upper limit of normal [ULN])
* History of gall bladder abnormalities
* History of any endocrine disorder
* History of alcohol or substance abuse within 2 years prior to Screening
* Positive urine screen for drugs of abuse and cotinine
* Consumption of caffeine- and/or xanthine containing products (eg, cola, coffee, tea, chocolate) within 72 hours prior to Check-in
* Consumption of alcohol within 48 hours prior to Check in
* Consumption of grapefruit, Seville oranges, and grapefruit- or Seville orange containing products within 72 hours prior to Check in

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of telotristat ethyl | Days 1, 2, 3, 6, 7, 8
Plasma concentrations of metabolite LP-778902 | Days 1, 2, 3, 6, 7, 8

SECONDARY OUTCOMES:
Number of treatment-emergent adverse events | Up to 39 days

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Daytona Beach, Florida, United States